CLINICAL TRIAL: NCT02177890
Title: Effect of Transcutaneous Vagal Nerve Stimulation on Reducing Visually Induced Motion Sickness in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wingate Institute of Neurogastroenterology (Other)
Responsible Party: Principal Investigator, Adam Farmer, Research fellow, Wingate Institute of Neurogastroenterology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-Farmer
Record Dates: First submitted 2014-06-24; First posted 2014-06-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Visually Induced Motion Sickness in Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcutaneous vagal nerve stimulation (Experimental): Active vagal nerve stimulation to the left auricular branch of the vagus nerve
  Interventions: Device: Transcutaneous vagal nerve stimulation
- Sham vagal nerve stimulation (Placebo Comparator): Placebo vagal nerve stimulation - stimulator attached to the ear but rotated 180 degrees so that it is not stimulating the vagus nerve.
  Interventions: Device: Sham vagal nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation
  Other Names: NEMOS
  Arms: Transcutaneous vagal nerve stimulation
Device: Sham vagal nerve stimulation
  Arms: Sham vagal nerve stimulation

SUMMARY:
Nausea is a common and distressing experience that often precedes vomiting. Amongst symptoms emanating from the gastrointestinal (GI) tract nausea can be considered somewhat unique, as on one hand it represents a normal, highly conserved, physiological response to an ingested toxin yet on the other it may indicate pathology. Nausea may also arise as a consequence of pharmaco- and chemotherapeutic interventions. Nausea negatively impacts on quality of life, adherence to treatment and is a cause for discontinuation of the development of novel compounds. Experimentally, nausea can be induced in humans using a visually induced motion stimulus. Previously we have developed a 10-minute motion video of the landscape rotating as seen from the perspective of a subject standing on Westminster Bridge, London. The tilted and rotating view visual display makes the subject perceive that they are spinning round and round on a spot tilted away from centre of gravity due to circular vection. This motion video induced nausea in approximately 50% of healthy participants and caused a reduction in cardiac vagal tone, a validated measure of the parasympathetic nervous system branch on the autonomic nervous system. We therefore are evaluating the role of external transcutaneous vagal nerve stimulation in visually induced motion sickness.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, aged 18-65, from staff, students and local population of Queen Mary, University of London.
2. Inclusion will be determined on the basis of availability, with no prior selection bias included. They should be able to attend the Wingate Institute for at least 2 x 1 hour sessions.
3. Subjects who score >15 on MSSQ (suggesting that they are sensitive to visually induced nausea).

Exclusion Criteria:

1. Subjects unable to provide informed consent.
2. Subjects with any systemic disease or medications that may influence the autonomic nervous system (e.g. beta-agonists or Parkinson's disease).
3. Subjects who score <15 on MSSQ (suggesting that they are insensitive to visually induced nausea).
4. Pregnant females to prevent any confounding effects on pregnancy related nausea.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Reduction of the subjective sensation of nausea on a visual analogue scale | 10 minutes

SECONDARY OUTCOMES:
Effect of transcutaneous vagal nerve stimulation on cardiac vagal tone | 10 minutes
Tolerability of transcutaneous vagal nerve stimulation | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Adam D Farmer, PhD MRCP, Principal Investigator — Wingate Institute
Locations (1):
- Wingate Institute of Neurogastroenterology, London, London, United Kingdom

REFERENCES:
- [Background] Farmer AD, Al Omran Y, Aziz Q, Andrews PL. The role of the parasympathetic nervous system in visually induced motion sickness: systematic review and meta-analysis. Exp Brain Res. 2014 Aug;232(8):2665-73. doi: 10.1007/s00221-014-3964-3. Epub 2014 May 4. PMID 24792503
- See also: Vagal nerve stimulator information — http://www.cerbomed.com/